CLINICAL TRIAL: NCT03733327
Title: Busulfan+ Cyclophosphamide+ Etoposide Conditioning Regimen for Primary Central Nervous System Lymphoma Undergoing Autologous Hematopoietic Stem Cell Transplantation
Brief Title: BUCYE Conditioning Regimen for PCNSL Undergoing Auto-HSCT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Peking University People's Hospital (Other); Guangzhou First People's Hospital (Other); Zhujiang Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Qifa Liu, Prof., Nanfang Hospital, Southern Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BUCYE-PCNSL-2018
Record Dates: First submitted 2018-11-06; First posted 2018-11-07 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Primary Central Nervous System Lymphoma; Autologous Hematopoietic Stem Cell Transplantation; Conditioning
MeSH Terms: interventions — Busulfan; Cyclophosphamide; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BUCYE (Experimental): For PCNSL patients undergoing auto-HSCT，BUCYE conditioning regimen was BU 3.2 mg/kg/day on days -7 and -4；CY 60 mg/kg/day on days -3 and -2; VP-16 15mg/kg/ day on days -3 and -2.
  Interventions: Drug: Busulfan (BU); Drug: Cyclophosphamide (CY); Drug: Etoposide (VP-16)

INTERVENTIONS:
Drug: Busulfan (BU) — Busulfan was administered at 3.2 mg/kg/day on days-7 to -4.
Drug: Cyclophosphamide (CY) — Cyclophosphamide was administered at 60 mg/kg/day on days -3 to -2.
Drug: Etoposide (VP-16) — Etoposide was administered at 15 mg/kg/day on days -3 to -2.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of BUCYE conditioning regimens in primary central nervous system lymphoma undergoing autologous hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
The prognosis of patients with primary central nervous system lymphoma (PCNSL) is poor. Recent studies have demonstrated that autologous hematopoietic stem cell transplantation (auto-HSCT) could improve the prognosis of these patients. However, the optimal conditioning regimen of auto-HSCT remains unclear. In this study, the investigators evaluated the safety and efficacy of BUCYE conditioning regimens in PCNSL undergoing auto-HSCT.

ELIGIBILITY:
Inclusion Criteria:

* Primary central nervous system lymphoma patients
* Achieving CR or PR, then mobilizing and collecting of peripheral blood stem cells

Exclusion Criteria:

* Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure)
* Patients with any conditions not suitable for the trial (investigators' decision)

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
OS | 2 year
  overall survival (OS)

SECONDARY OUTCOMES:
DFS | 2 year
  disease-free survival (DFS)
relapse rate | 2 year
  relapse rate
TRM | 2 year
  transplant-related mortality (TRM)

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided